CLINICAL TRIAL: NCT01232452
Title: An Open-label, Multicenter, Randomized Phase 2 Study Evaluating the Safety and Efficacy of Cisplatin and Pemetrexed With or Without Cixutumumab as First-Line Therapy in Patients With Advanced Nonsquamous Non-Small Cell Lung Carcinoma
Brief Title: A Study in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13973; I5A-MC-JAEM (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-28; First posted 2010-11-02 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: lung cancer; advanced; non-small cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed; Cisplatin; cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pemetrexed + Cisplatin + Cixutumumab (Experimental): Induction Treatment: Pemetrexed 500 mg/m^2 plus cisplatin 75 mg/m^2 plus cixutumumab 20 mg/kg given intravenously (IV) on Day 1 of a 21 day cycle for up to 4 cycles. Two additional cycles of cisplatin may be given (6 cycles total) for patients with significant tumor size reduction, after sponsor approval.
  Maintenance Therapy: Pemetrexed 500 mg/m^2 plus cixutumumab 20 mg/kg given IV every 21 days until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Cixutumumab
- Pemetrexed + Cisplatin (Active Comparator): Induction Treatment: Pemetrexed 500 mg/m^2 plus cisplatin 75 mg/m^2 given intravenously (IV) on Day 1 of a 21 day cycle for up to 4 cycles. Two additional cycles of cisplatin may be given (6 cycles total) for patients with significant tumor size reduction, after sponsor approval.
  Maintenance Therapy: Pemetrexed 500 mg/m^2 given IV every 21 days until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — Administered intravenously (IV)
  Other Names: Alimta; LY231514
Drug: Cisplatin — Administered IV
Drug: Cixutumumab — Administered IV
  Other Names: LY3012217
  Arms: Pemetrexed + Cisplatin + Cixutumumab

SUMMARY:
The primary purpose of this study is to evaluate the hypothesis that cixutumumab given in combination with cisplatin and pemetrexed is superior to cisplatin and pemetrexed as first-line therapy for patients with advanced nonsquamous non-small cell lung carcinoma (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed, nonsquamous (adenocarcinoma/large cell or other) NSCLC.
* The participant has Stage IV disease at the time of study entry.
* Participants with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, and stereotactic radiosurgery) ending at least 14 days prior to randomization, or after surgical resection performed at least 28 days prior to randomization. The participant may have no evidence of Grade 1 (or greater) Central Nervous System (CNS) hemorrhage based on pretreatment scans(performed within 21 days before randomization).
* The participant has measurable or nonmeasurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 guidelines.
* The participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* If prior adjuvant or neoadjuvant chemotherapy, the last dose of adjuvant or neoadjuvant treatment was administered at least 6 months prior to randomization.
* The participant has adequate bone marrow reserve, and renal and hepatic function
* The participant has fasting serum glucose less than or equal to 125 mg/dL, and hemoglobin A1C less than or equal to 6%.
* Females with reproductive potential: Must have a negative serum or urine pregnancy test within 7 days prior to the first dose of any study drug.
* Males and females with reproductive potential: Must agree to use medically approved contraceptive precautions during the study and for 6 months following the last dose of any study drug.
* The participant has the ability to understand and the willingness to sign a written informed consent form.
* Previous radiation therapy is allowed to less than 25% of the bone marrow, but should have been limited and must not have included whole pelvis radiation.
* The participant has archived tumor tissue available for analysis (can be either primary tumor or metastases).
* The participant has an estimated life expectancy of at least 12 weeks.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participants who have squamous histology.
* The participant's tumor fully or partially contains Small Cell Lung Cancer (SCLC).
* The participant has leptomeningeal disease.
* The participant is currently or has previously received chemotherapy for advanced (Stage IV) NSCLC.
* The participant has a history of treatment with other agents targeting the Insulin-like or Epidermal Growth factor receptors.
* Participants who have received prior Pemetrexed treatment.
* The patient has a known allergy/history of hypersensitivity reaction to any of the treatment components.
* The participant has diabetes mellitus as defined by being treated with glucose lowering medications in the past 3 months prior to enrollment.
* The participant has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, uncontrolled hypertension, clinically significant cardiac arrhythmia,or psychiatric/social situations that would limit compliance with study requirements.
* The participant has an ongoing or active infection requiring parenteral antibiotic, antifungal, or antiviral therapy.
* The participant has undergone major surgery within 28 days prior to randomization.
* The participant has received a prior autologous or allogeneic organ or tissue transplantation.
* The participant is pregnant or lactating.
* The participant has a history of another primary cancer, with the exception of the following: curatively resected nonmelanomatous skin cancer, curatively treated carcinoma in situ, or other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the last 5 years.
* The participant has superior vena cava syndrome contraindicating hydration.
* The participant has current clinically-relevant coronary artery disease (New York Heart Association III or IV) or uncontrolled congestive heart failure.
* The participant has any Grade 2 (or greater) peripheral neuropathy.
* The participant has clinically significant third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry.
* The participant is unable to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than an aspirin dose less than or equal to 1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* The participant is unwilling or unable to take premedications (folic acid, vitamin B12, or corticosteroids) required by the pemetrexed label.
* The participant has received a recent (within 30 days of enrollment) or is receiving concurrent yellow fever vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hackensack, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Argentina (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rioja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendoza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Fe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viedma
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duffel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Brazil (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barretos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ijuí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salvador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São José do Rio Preto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oshawa, Ontario, Canada
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clermont-Ferrand
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Braunschweig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beer Yaakov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perugia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saronno
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harderwijk
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Girona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edirne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zeytinburnu

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are those participants who died or had progressive disease (PD).
Groups:
- Pemetrexed + Cisplatin + Cixutumumab: Induction Treatment: Pemetrexed 500 mg/m^2 plus cisplatin 75 mg/m^2 plus cixutumumab 20 mg/kg given intravenously (IV) on Day 1 of a 21 day cycle for up to 4 cycles. Two additional cycles of cisplatin may be given (6 cycles total) for participants with significant tumor size reduction, after sponsor approval.
  Maintenance Therapy: Pemetrexed 500 mg/m^2 plus cixutumumab 20 mg/kg given IV every 21 days until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
- Pemetrexed + Cisplatin: Induction Treatment: Pemetrexed 500 mg/m^2 plus cisplatin 75 mg/m^2 given IV on Day 1 of a 21 day cycle for up to 4 cycles. Two additional cycles of cisplatin may be given (6 cycles total) for participants with significant tumor size reduction, after sponsor approval.
  Maintenance Therapy: Pemetrexed 500 mg/m^2 given IV every 21 days until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Started | 87 | 85
Received at Least One Dose of Study Drug | 85 | 81
Completed | 48 | 46
Not Completed | 39 | 39
Not completed — Adverse Event | 17 | 15
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Physician Decision | 8 | 12
Not completed — Protocol entry criterion not met | 0 | 2
Not completed — Sponsor Decision | 3 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed + Cisplatin + Cixutumumab: Induction Treatment: Pemetrexed 500 mg/m^2 plus cisplatin 75 mg/m^2 plus cixutumumab 20 mg/kg given IV on Day 1 of a 21 day cycle for up to 4 cycles. Two additional cycles of cisplatin may be given (6 cycles total) for participants with significant tumor size reduction, after sponsor approval.
  Maintenance Therapy: Pemetrexed 500 mg/m^2 plus cixutumumab 20 mg/kg given IV every 21 days until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin | Total
Number analyzed (Participants) | 87 | 85 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.87) | 59.3 (9.96) | 59.4 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 54 | 53 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 24 | 37
  Not Hispanic or Latino | 45 | 33 | 78
  Unknown or Not Reported | 29 | 28 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 81 | 80 | 161
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants] — Population: All randomized participants who received one dose of study drug and had evaluable Region of Enrollment data.
  Participants
    Canada: number analyzed (Participants) | 1 | 1 | 2
    Canada | 1 | 1 | 2
    Netherlands: number analyzed (Participants) | 4 | 1 | 5
    Netherlands | 4 | 1 | 5
    Argentina: number analyzed (Participants) | 5 | 8 | 13
    Argentina | 5 | 8 | 13
    Turkey: number analyzed (Participants) | 5 | 7 | 12
    Turkey | 5 | 7 | 12
    Belgium: number analyzed (Participants) | 7 | 6 | 13
    Belgium | 7 | 6 | 13
    United States: number analyzed (Participants) | 9 | 11 | 20
    United States | 9 | 11 | 20
    Brazil: number analyzed (Participants) | 13 | 21 | 34
    Brazil | 13 | 21 | 34
    Italy: number analyzed (Participants) | 9 | 8 | 17
    Italy | 9 | 8 | 17
    Israel: number analyzed (Participants) | 6 | 2 | 8
    Israel | 6 | 2 | 8
    France: number analyzed (Participants) | 3 | 2 | 5
    France | 3 | 2 | 5
    Germany: number analyzed (Participants) | 17 | 8 | 25
    Germany | 17 | 8 | 25
    Spain: number analyzed (Participants) | 6 | 6 | 12
    Spain | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from date of randomization until the date of disease progression, or death from any cause, whichever was first. Disease progression was assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, and/or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions. Participants without documentation for disease progression or death were censored at the date of last tumor assessment. The PFS was estimated following the Kaplan-Meier method.
Time Frame: Randomization Date to Disease Progression or Death From Any Cause Up to 18.3 Months
Population: All randomized participants. Participants censored in Cixutumumab arm = 20 and Pemetrexed + Cisplatin arm = 21.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Number analyzed (Participants) | 87 | 85
months | 5.45 [3.88 to 6.05] | 5.22 [4.24 to 6.74]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin + Cixutumumab vs Pemetrexed + Cisplatin; Test type: Superiority; p = 0.848, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.73 to 1.47]

2. Secondary Outcome: Percentage of Participants Achieving an Objective Response Rate (ORR)
Description: The ORR is the percentage of all participants with Partial Response (PR) or Complete Response (CR) according to RECIST v1.1. Disease progression was defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, and/or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions. ORR is confirmed best overall tumor response of CR and PR. CR was defined as the disappearance of all target and non-target lesions; PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD.
Time Frame: Randomization to Disease Progression Up to 18.3 Months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Number analyzed (Participants) | 87 | 85
percentage of participants | 37.9 [27.7 to 49.0] | 30.6 [21.0 to 41.5]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin + Cixutumumab vs Pemetrexed + Cisplatin; Test type: Superiority; p = 0.338, Fisher Exact

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death from any cause. If the participant is alive at the end of the follow-up period or is lost to follow-up, OS will be censored on the last date the participant is known to be alive. OS was estimated using the Kaplan-Meier method.
Time Frame: Randomization Date to Death From Any Cause Up to 20 Months
Population: All randomized participants. Participants censored cixutumumab arm = 47 and pemetrexed + cisplatin arm = 39.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Number analyzed (Participants) | 87 | 85
Months | 10.68 [8.74 to NA] — The upper limit was not estimable due to the data had insufficient overall survival data events. | 10.38 [7.43 to 14.39]

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that the criteria for PD is met, or death, is objectively documented. DOR was estimated using the Kaplan-Meier method. Disease progression was assessed via RECIST version 1.1, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, and/or the appearance of one or more new lesion(s), and/or unequivocal progression of existing non-target lesions
Time Frame: Time from Response to Disease Progression or Death from Any Cause Up to 20 Months
Population: All randomized participants who had CR or PR. Participants censored in Cixutumumab arm = 10 and Pemetrexed + Cisplatin arm = 8.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Number analyzed (Participants) | 33 | 26
Months | 4.90 [4.17 to 6.28] | 3.91 [2.92 to 6.41]

5. Secondary Outcome: Time to Progressive Disease (TTPS)
Description: TTPS was defined as the time from the date of randomization until the date of disease progression. Disease progression was assessed via RECIST version 1.1, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, and/or the appearance of one or more new lesion(s), and/or unequivocal progression of existing non-target lesions.TTPS was estimated using the Kaplan-Meier method.
Time Frame: Randomization Date to Disease Progression Up to 18.3 Months
Population: All randomized participants. Participants censored in Cixutumumab arm = 39 and in the Pemetrexed + Cisplatin arm = 36.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Number analyzed (Participants) | 87 | 85
Months | 6.05 [5.32 to 7.79] | 6.05 [4.93 to 7.89]

6. Secondary Outcome: Time to Worsening of Symptoms as Measured by Lung Cancer Symptom Scale (LCSS) Score
Description: TTPS was defined as the time from the date of randomization until the date of worsening of symptoms as measured by Lung Cancer Symptom Scale (LCSS) score. Symptomatic progression was defined as an increase (worsening) of the Average Symptomatic Burden Index (ASBI) that is, the mean of the six major lung cancer specific symptom scores of the LCSS patient scale - ranging from 0 to 100 where higher score indicates worst outcome). For each participant, the maximum improvement over baseline score was calculated for each of the 9 LCSS items, ASBI and LCSS total score. Participants without event are censored at the date of the last LCSS assessment. TTPS was estimated using the Kaplan-Meier method.
Time Frame: Time to worsening of symptoms as measured by LCSS score Up to 18.3 Months
Population: All randomized participants. Participants censored in Cixutumumab arm = 38 and Pemetrexed + Cisplatin arm = 46.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Number analyzed (Participants) | 87 | 85
Months | 2.14 [1.54 to 2.99] | 4.21 [2.43 to 5.36]

7. Secondary Outcome: Change in Tumor Size (CTS)
Description: CTS was measured by percentage change of tumor size at the end of Cycle 2 comparing to baseline tumor size.
Time Frame: Change from baseline measurement to the end of Cycle 2, average of 42 days
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Number analyzed (Participants) | 87 | 85
Percent Change | -23.88 (18.859) | -16.04 (26.143)

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Cixutumumab, Cycle 1 (First Infusion) and Cycle 4 (Fourth Infusion)
Time Frame: First Infusion: [Prior to Infusion (of Cycle1): 1, 72, 168, 336 hours(hrs) and 504 hrs (i.e. Prior to Infusion of Cycle 2)] and Fourth Infusion; [Prior to Infusion (of Cycle 4),1,24,72,120,168,240,336 hrs and 504 hrs (i.e. Prior to Infusion of Cycle 5)]
Population: Participants who were randomized to the cixutumumab arm and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab
Number analyzed (Participants) | 71
microgram/milliliter (ug/mL)
  First Infusion | 481 (33)
  Fourth Infusion: number analyzed (Participants) | 31
  Fourth Infusion | 556 (17)

9. Secondary Outcome: PK: Area Under the Concentration Time Curve (AUC[0-inf]) of Cixutumumab, Cycle 1 (i.e. First Infusion)
Time Frame: Prior to Infusion (of Cycle 1), 1, 72, 168, 336 hrs and 504 hrs (i.e. Prior to Infusion of Cycle 2)
Population: Participants who were randomized to the cixutumumab arm and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (ug*hr/mL)
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab
Number analyzed (Participants) | 57
microgram*hour/milliliter (ug*hr/mL) | 73200 (35)

10. Secondary Outcome: PK: Area Under the Concentration Time Curve During 1 Dosing Interval (i.e. 504 hr, AUC(0-tau) of Cixutumumab, Cycle 4 (i.e. Fourth Infusion)
Time Frame: Prior to Infusion (of Cycle 4), 1, 24, 72, 120, 168, 240, 336 hrs and 504 hrs (i.e. Prior to Infusion of Cycle 5)
Population: Participants who were randomized to the cixutumumab arm and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ug*hr/mL)
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab
Number analyzed (Participants) | 27
(ug*hr/mL) | 79700 (30)

11. Secondary Outcome: Pharmacodynamics (PD) Markers: Free Insulin-like Growth Factor-I (IGF-I, Total IGF-I, and IGF Binding Proteins (IGFBP-3)
Description: Blood samples for the determination of PD marker concentrations were collected at the specified time points for all participants. Analysis of the following markers include free IGF-I, total IGF-I, and IGFBP-3.
Time Frame: Preinfusion, Cycle 2, Cycle 4, Cycle 8, Postinfusion, 30-Day Follow-Up
Population: Zero participants were analyzed for PD Biomarker IGF-I, total IGF-I, and IGFBP-3 due to blood samples were not collected in order to assess biomarker data.
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Immunogenicity of Cixutumumab
Time Frame: Preinfusion, Cycle1(C1): 1, 72, 168, 240, 336 hours(hrs); C2 and C3: 1, 168, 336 hrs; C4: 1, 24,72,120,168, 240, 336, 504 hrs, Postinfusion; 30 Day Follow Up
Population: Zero participants were analyzed due to no immunogenicity analysis was done and the assay was never developed.
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: 6 participants did not receive study drug after randomization. 2 of the participants were in the cixutumumab arm and 4 of the participants were in the control arm.
Arm/Group | Pemetrexed + Cisplatin + Cixutumumab | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 49/85 | 31/81
Other Adverse Events (participants affected / at risk) | 83/85 | 79/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin + Cixutumumab (N=85) | Pemetrexed + Cisplatin (N=81)
Anaemia (Blood and lymphatic system disorders) | 6 (18) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (3)
Pancytopenia (Blood and lymphatic system disorders) | 2 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (9) | 1 (1)
Fatigue (General disorders) | 7 (9) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 3 (4)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 1 (2) | 4 (7)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (7) | 0 (0)
White blood cell count decreased (Investigations) | 2 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (3)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Osteosynthesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (4) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin + Cixutumumab (N=85) | Pemetrexed + Cisplatin (N=81)
Anaemia (Blood and lymphatic system disorders) | 33 (103) | 36 (98)
Leukopenia (Blood and lymphatic system disorders) | 6 (12) | 5 (27)
Neutropenia (Blood and lymphatic system disorders) | 12 (29) | 17 (35)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (31) | 5 (9)
Vertigo (Ear and labyrinth disorders) | 9 (11) | 4 (4)
Lacrimation increased (Eye disorders) | 8 (8) | 7 (10)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 11 (15)
Constipation (Gastrointestinal disorders) | 27 (39) | 19 (28)
Diarrhoea (Gastrointestinal disorders) | 19 (29) | 16 (21)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 45 (74) | 41 (101)
Stomatitis (Gastrointestinal disorders) | 14 (24) | 6 (8)
Vomiting (Gastrointestinal disorders) | 29 (41) | 28 (55)
Asthenia (General disorders) | 10 (12) | 9 (30)
Chest pain (General disorders) | 2 (3) | 5 (10)
Fatigue (General disorders) | 36 (82) | 33 (63)
Influenza like illness (General disorders) | 1 (1) | 6 (7)
Mucosal inflammation (General disorders) | 12 (18) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (4) | 6 (6)
Oedema peripheral (General disorders) | 7 (7) | 13 (19)
Pyrexia (General disorders) | 5 (5) | 10 (14)
Conjunctivitis (Infections and infestations) | 3 (5) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (7)
Alanine aminotransferase increased (Investigations) | 8 (11) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 5 (7)
Blood creatinine increased (Investigations) | 12 (18) | 16 (20)
Neutrophil count decreased (Investigations) | 9 (24) | 6 (10)
Platelet count decreased (Investigations) | 6 (6) | 9 (14)
Weight decreased (Investigations) | 17 (28) | 11 (13)
White blood cell count decreased (Investigations) | 5 (10) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 24 (36) | 27 (32)
Dehydration (Metabolism and nutrition disorders) | 10 (13) | 6 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 43 (156) | 16 (45)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (8) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (7) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (13) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 10 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Dizziness (Nervous system disorders) | 11 (13) | 5 (7)
Dysgeusia (Nervous system disorders) | 7 (9) | 8 (10)
Paraesthesia (Nervous system disorders) | 2 (3) | 5 (5)
Anxiety (Psychiatric disorders) | 3 (3) | 5 (6)
Depression (Psychiatric disorders) | 5 (5) | 4 (4)
Insomnia (Psychiatric disorders) | 5 (5) | 7 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (21) | 16 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (21) | 16 (26)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (5)
Hypotension (Vascular disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days